CLINICAL TRIAL: NCT04553198
Title: Quantifying the Role of Sensory Systems Processing in Post-Stroke Walking Recovery
Acronym: BLT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: American Academy of Neurology (Other)
Responsible Party: Principal Investigator, Oluwole Awosika, MD, MSCR, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0450
Record Dates: First submitted 2020-09-06; First posted 2020-09-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Chronic Stroke; Walking, Difficulty; Gait, Hemiplegic
Keywords: Gait; Balance; Non-body weight supported treadmill training; Backward locomotion treadmill training; Forward locomotion treadmill training; Walking Rehabilitation; Walking Recovery
MeSH Terms: conditions — Stroke; Mobility Limitation; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: stratified randomization
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is blinded to the intervention type.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backward Locomotion Treadmill Training (BLTT) (Experimental): Participants train on a reverse treadmill (no bodyweight support), three times per week x 3 weeks.
  Interventions: Behavioral: Backward Locomotion Treadmill Training (BLTT)
- Forward Locomotion Treadmill Training (FLTT) (Sham Comparator): Participants train on a treadmill (no bodyweight support), three times per week x 3 weeks.
  Interventions: Behavioral: Backward Locomotion Treadmill Training (BLTT)

INTERVENTIONS:
Behavioral: Backward Locomotion Treadmill Training (BLTT) — 9-training sessions of reverse treadmill training (no bodyweight support)over three weeks.

SUMMARY:
Despite current walking rehabilitation strategies, the majority of stroke survivors are unable to walking independently in the community and remain at increased risk of falls. Backward treadmill training is a novel training approach used by elite athletes to enhance speed, agility, and balance; however, it is currently unknown how this exercise interacts with the central nervous system or if it could benefit stroke survivors with residual walking impairment. Knowledge gained from this study will likely lead to more effective walking rehabilitation strategies in stroke and related disorders.

DETAILED DESCRIPTION:
Walking impairment after a stroke impacts nearly 66% of stroke survivors and is a rising cause of morbidity worldwide. Despite ongoing efforts to increase the quality and delivery of rehabilitative care, less than ten percent of stroke survivors ever achieve walking independence within the community and are at higher risk of falls, fractures, rehospitalization. Several factors may lead to walking impairment, but the two most prevalent causes are lower extremity asymmetry and imbalance. Herein, the investigators propose backward locomotion treadmill training (BLTT), as a promising approach for walking rehabilitation in stroke survivors.

Hence, our central hypothesis is that BLTT facilitates sensory signaling, leading to an improvement in walking speed. The investigators have preliminary proof of technique and feasibility data suggesting that BLTT is safe and feasible for stroke patients, with our results showing clinically meaningful improvement in overground walking speed after just six training sessions, with retention at the two-week follow-up. The next logical step in planning toward a future definitive clinical trial is to determine its preliminary efficacy compared with conventional forward walking treadmill training (FLTT) as control.

The investigators plan to test the preliminary efficacy of BLTT by conducting a prospective, randomized, blinded-endpoint, pilot study of 40 individuals with residual mild-moderate gait impairment, >6 months post-stroke, to BLTT (n=20) versus FLTT (n=20), for nine 30-minute training session (3 sessions/week). The investigators will utilize well-validated behavioral measures in stroke recovery and rehabilitation to test the following Aims:

Aim 1. Determine the training-related effects of BLTT on overground walking speed (primary outcome) To achieve this aim, the investigators will compare the Pre-Post change in walking speed [10- meter walk test (10MWT)] between groups. Our working hypothesis 1 is that BLTT will increase walking speed (>0.13m/s), compared to the control group (FLTT).

Aim 2. Determine the effects of training on walking symmetry, proprioceptive signaling, and dynamic balance. The Zeno Walkway Gait Analysis software will capture Pre-Post changes in temporal gait symmetry index during the 10-MWT. Working hypothesis 2a: BLTT will be associated with a favorable improvement in the temporal symmetry index score. Proprioception and spinovestibular function will be measured with the modified Sensorineural Integration Test (mSIT), and dynamic balance will be assessed with the completion time on the instrumented Timed Up & Go (i-TUG). Working hypothesis 2b and c: BLTT will be associated with a favorable improvement Pre-Post mSIT(b) and completion time on the i-TUG (c).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Ability to maintain ≥0.3mph speed for 6-minute interval on the treadmill
* Able to walk independently (cane and hemi-walker acceptable)
* Ambulate >10 meters over ground with the Free Step Harness System (as a safety precaution)
* Discharged from formal rehabilitation.

Exclusion Criteria:

* Walking speed <0.4m/s (per 10MWT comfortable)
* Unstable cardiac status which would preclude participation in a moderate-intensity exercise program
* Significant language barrier which might prevent the participant from following instructions during training and testing
* Adverse health condition that might affect walking capacity (severe arthritis, significant pulmonary disease significant ataxia, or severe hemi-neglect)
* Severe lower extremity spasticity (Ashworth >2)
* Depression (>10 on the Patient Health Questionnaire, if untreated).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Change in 10-Meter Walk (fast) | Pre-Baseline (Day of Randomization) to One Day Post-Training
  Two 10MWT trials (using a stop-watch) are averaged and documented in meters/second.

SECONDARY OUTCOMES:
10-Meter Walk Test (Fast- Retention) | One Day Post Training, One month Post Training, 3- Months Post Training
  Two 10MWT (fast) trials (using a stop-watch) are averaged and documented in meters/second.
10-Meter Walk (Comfortable) | Baseline (Day of Randomization), One Day Post-Training, One month Post Training, 3-Months Post Training
  wo 10MWT trials (using a stop-watch) are averaged and documented in meters/second.

OTHER OUTCOMES:
Temporal Symmetry Index | Baseline (Day of Randomization), One Day Post-Training, One month Post Training, 3- Months Post Training
  %-limb support of the affected and unaffected leg, during the 10 MWT
Static Balance: Sway Index (SI) | Baseline (Day of Randomization), One Day Post-Training, One month Post Training, 3- Months Post Training
  The Biodex Modified Clinical Test of Sensory Interaction on Balance (mSIBT) is a well-validated balance system and has been used neurally intact and neurologically impaired individuals to objectively measure static balance. Compared to other measures of static balance, the mSIBT provides the added benefit of differentiating the contributions of the visual, proprioceptive and vestibular systems. Method: While on the platform (with safety harness), participants will stand with the hands at the side under 4 conditions (30 secs/condition):1) firm surface with the eyes open, 2) firm surface with the eyes closed, 3) compliant surface (foam) with the eyes open, 4) Compliant surface (foam) with the eyes closed. Three attempts will be average and documented as SI.
Dynamic Balance: Instrumented Timed Up & Go (i-TUG)- 3 Meter | Baseline, One Day Post-Training, One month Post Training, 3- Months Post Training
  Participants will be instructed to sit with the back against the chair (seat height 46cm, arm height 67cm) and on the word "go," stand up, walk at a comfortable speed past the 3-m mark, turn around, walk back, and sit down in the chair. Two trials are averaged and documented in seconds.
Dynamic Balance: Instrumented Timed Up & Go (i-TUG)- 7 Meter | Baseline, One Day Post-Training, One month Post Training, 3- Months Post Training
  Participants will be instructed to sit with the back against the chair (seat height 46cm, arm height 67cm) and on the word "go," stand up, walk at a comfortable speed past the 7-m mark, turn around, walk back, and sit down in the chair. Two trials are averaged and documented in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No